CLINICAL TRIAL: NCT01253785
Title: Pulse Oximeter Responses to Multiple Levels of Stable Hypoxia
Status: Completed | Type: Observational
Sponsor: SterilMed, Inc. (Industry)
Responsible Party: Garrett Ahlborg, SterilMed, Inc.
Other Study IDs: STER05
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Validate pulse oximeter sensor SpO2 accuracy from 70-100% during induced hypoxia.

DETAILED DESCRIPTION:
The testing is conducted on 10 healthy, consenting, non-smoking subjects in accordance with the IRB approved Protocol. The subjects shall be distributed across both genders and a range of skin tones as equally as practical.

An arterial line will be placed in the radial artery of each subject's right arm, and sensors will be attached to each subject. The subjects will be placed in a semi-supine position and allowed to breathe through a mouthpiece while the nose is blocked with a nose-clip.

Hypoxia will be induced by on each subject, as levels of oxyhemoglobin saturation (between 70% and 100%) are achieved by breathing mixtures of nitrogen, room air and carbon dioxide. Inspired O2 concentration will be adjusted breath-by-breath using a computed saturation, based on end-tidal PO2 and PCO2, as sampled by a mass spectrometer. Predicted levels of oxyhemoglobin saturations will be attained and held stable. At a minimum of sixty seconds into each plateau, a 0.5cc waste blood draw through the arterial line, followed by the first 1.0cc sample blood draw. After approximately thirty additional seconds, the second 1.0cc sample blood draw will be taken. The samples will immediately be analyzed by a Radiometer OSM-3 multi-wavelength co-oximeter and recorded. The SpO2 data from the oximeters will be collected via a laptop computer. Concurrent with the end of each blood draw, a marker will be generated on the laptop computers to identify the event.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* 18 years or older
* Meet the requirements of the investigator's medical history questionnaire criteria which described family history, present symptoms, smoking history, risk factors, nutrition, exercise levels and stress levels
* Understand and provide signed consent for the procedure

Exclusion Criteria:

* Smoker
* User of illegal drugs
* Hypertension
* Respiratory disease
* Known allergy to Lidocaine or its derivatives
* Those suffering from upper respiratory infection on the day of study

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, consenting, non-smoking subjects, 18 years or older, both genders and a range of skin tones.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
SpO2 Accuracy Verification Study (Arms) of ≤ 3.0% between 70-100% | During Analysis - data were collected for all subjects on one day

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E Bickler, MD, PhD, Principal Investigator — University of California, San Francisco